CLINICAL TRIAL: NCT00872625
Title: Phase I Study - Hypofractionated Cyberknife Radiotherapy Combined With Neoadjuvant Chemotherapy for Breast Tumors
Brief Title: Radiation Therapy and Docetaxel Followed by Standard Therapy in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/24; CALACASS-CYBERNEO; CALACASS-2006/24; INCA-RECF0621; 2006-A00250-51 (Other: AFSSAPS ID RCB)
Record Dates: First submitted 2009-03-28; First posted 2009-03-31 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2015-02

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Neoadjuvant Therapy; Radiotherapy, Image-Guided; Radiotherapy; Radiosurgery

ARMS (1):
- Cyberknife (Experimental)
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: epirubicin hydrochloride; Drug: fluorouracil; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: hypofractionated radiation therapy; Radiation: image-guided radiation therapy; Radiation: radiation therapy; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: hypofractionated radiation therapy
Radiation: image-guided radiation therapy
Radiation: radiation therapy
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in higher doses over a shorter period of time may kill more tumor cells and have fewer side effects. Drugs used in chemotherapy, such as docetaxel, epirubicin, cyclophosphamide, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of radiation therapy when given together with docetaxel followed by standard therapy in treating women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tolerance to concurrent neoadjuvant docetaxel and cyberknife hypofractionated radiotherapy followed by standard treatment in women with breast cancer in order to find the maximum-tolerated dose of radiotherapy.

Secondary

* Evaluate the efficacy of the combination chemoradiotherapy.
* Evaluate breast-conserving surgery.
* Evaluate the quality of life.

OUTLINE: This is a dose-escalation study of cyberknife hypofractionated radiotherapy.

Patients receive neoadjuvant docetaxel IV on day 1. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Beginning during the first or second course of neoadjuvant chemotherapy, patients undergo hypofractionated radiotherapy. Patients then receive standard chemotherapy comprising epirubicin hydrochloride IV, cyclophosphamide IV, and fluorouracil IV on day 1. Treatment repeats every 3 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients undergo surgery 4-8 weeks after the last course of chemotherapy, and then undergo standard radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of breast cancer

  * Unifocal disease
  * Non-metastatic disease
  * Not a candidate for breast-conserving surgery
* No superficial breast cancer (defined as the distance between tumor and skin ≤ 1 cm)
* Undergone MRI of the breast to define the macroscopic tumor volume
* Undergone scanning of the breast to mark the location for radiotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No counter-indications to surgery, standard neoadjuvant chemotherapy, or insertion of an implantable venous device
* No patient for whom clinical follow up is impossible for psychological, familial, social, or geographical reasons
* No patients deprived of liberty or under trusteeship

PRIOR CONCURRENT THERAPY:

* No prior ipsilateral breast irradiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of radiotherapy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Bondiau, MD, PhD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France